CLINICAL TRIAL: NCT04729868
Title: Ultrasound Guided Infraclavicular Brachial Plexus Block Using Levo-bupivacaine Alone or Combined With Dexmedetomidine for Hand and Forearm Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Zaher Zaki Zaher, director, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: aswu/125/4/17
Record Dates: First submitted 2021-01-07; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Acquired Deformity of Elbow; Forearm; Hand; Wrist

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group Levo-bupivacaine (Other): Group A (20 patients): Anesthesia will be performed with 35 ml of 0.5% levo-bupivacaine plus 1ml normal saline under the guidance of ultrasound for infraclavicular brachial plexus block.
  Interventions: Drug: Levobupivacaine(chirocaine) plus dexmedetomidine(precedex)
- group levo-bupivacaine plus 50µg dexmedetomidine (Other): Group B (20 patients): Anesthesia will be performed with 35 ml of 0.5% levo-bupivacaine plus 50µg dexmedetomidine under the guidance of ultrasound for infraclavicular brachial plexus block.
  Interventions: Drug: Levobupivacaine(chirocaine) plus dexmedetomidine(precedex)
- group levo-bupivacaine plus 100µg dexmedetomidine (Other): Group C (20 patients): Anesthesia will be performed with 35 ml of 0.5% levo-bupivacaine plus 100µg dexmedetomidine under the guidance of ultrasound for infraclavicular brachial plexus block.
  Interventions: Drug: Levobupivacaine(chirocaine) plus dexmedetomidine(precedex)

INTERVENTIONS:
Drug: Levobupivacaine(chirocaine) plus dexmedetomidine(precedex) — evaluate the efficacy of levo-bupivacaine alone and with dexmedetomidine in Ultrasound guided infraclavicular brachial plexus block for hand and forearm surgeries
  Other Names: the efficacy of levo-bupivacaine alone and with dexmedetomidine in Ultrasound guided infraclavicular brachial plexus block for hand and forearm surgeries

SUMMARY:
To evaluate the efficacy of levo-bupivacaine alone and with dexmedetomidine in Ultrasound guided infraclavicular brachial plexus block for hand and forearm surgeries as regard:

Onset of sensory and motor blockade. Duration of sensory and motor blockade.

Analgesic pain scores using the verbal rating scale (VRS) for pain. Duration of analgesia postoperative complications.

DETAILED DESCRIPTION:
Technique for ultrasound guided infraclavicular brachial plexus block:

Preliminary scan

* The patient is positioned supine with the arm abducted to 90°(or resting by their side if unable to do so).
* The probe is placed immediately medial to the coracoid process in the parasagittal plane.
* Identify the pectoralis major and minor muscles superficially and the axillary artery and vein(s) deep to this. The vein is usually caudad relative to the artery.
* The cords of the brachial plexus are seen as either hypoechoic or hyperechoic structures positioned around the axillary artery. The lateral cord is lateral (cephalad) to the artery, the medial cord medial (caudad),and the posterior cord posterior (deep). They can be difficult to visualize but are usually positioned closely to the artery.

Ultrasound settings

* Probe: high-frequency (>10MHz) linear broadband probe.
* Settings: MB-resolution/general.
* Depth: 3-6cm.
* Orientation: parasagittal.
* Needle: 50-100mm depending on depth of plexus. Technique
* An in-plane approach is recommended, inserted from the cephalad end of the transducer.
* Needle tip visualization may be challenging as the needle angle can be quite steep.
* Prepare the skin with 0.5% chlorhexidine in 70% alcohol. Wait until the skin is dry.
* Anaesthetize the skin with a subcutaneous injection of 1% lidocaine at the point of needle insertion.
* The needle is first advanced posterolateral to the artery to deposit local anesthetic around the posterior cord, 5 o'clock position on artery.
* After careful aspiration LA is injected in small aliquots, observing the spread of the LA which ideally occurs behind and up both sides of the artery forming a 'U' shape around the artery, 1-9 o'clock around the artery.
* If medial (caudad) spread is not observed then reinsertion of the needle between the axillary artery and vein, adjacent to the medial cord may be required.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-65 years old.
* American society of anesthesiologist physical status (ASA): I-II.
* Operation: forearm & hand surgeries.

Exclusion Criteria:

* Patients with chronic pain
* Those using chronic analgesic medications
* History of brachial plexus injury
* Allergy to the study drugs
* Hepatic or renal insufficiency or infection at the site of injection

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Onset time of sensory block in minutes | 45 minutes
  After the injection of the solution, every patient was checked for the onset of sensory blockade using goose soaked with iced normal saline by the following scale (three-point scale): Grade 0= perceived as normal sensation, Grade 1 = loss of cold sensation (analgesia), Grade 2= loss of sensation of touch (anesthesia).
onset time of motor blockade in minutes using the modified Bromage scale (Three-point scale) | 24 hours
  the modified Bromage scale (Three-point scale): Grade 0: Normal motor function, Grade 1: Decreased motor strength with the ability to move the fingers only, Grade 2: Complete motor block with an inability to move the fingers.
Duration of sensory block in hours | 24 hours
  It's the time from sensory block onset to the time of restoration of sensation at the surgical site
Duration of motor block in hours | 24 hours
  It's the time from motor block onset to the restoration of global mobility in the hand and the wrist.

SECONDARY OUTCOMES:
Visual analog scale (VAS) | 24 hours
  the VAS consisted of a straight, vertical 10-cm line; the bottom point represented "no pain" = (0 cm) and the top "the worst pain you ever have" = (10 cm)
Postoperative first analgesic request time in hours | 24 hours
  was taken from the time of complete sensory block to the request to rescue analgesia when VAS > 4 cm.
Mean blood pressure in mmHg | 24 hours
  was measured before the block (0 min) and at 5, 10, 15, 30 min then 1, 2, 3, 6, 12,18and 24 h after the block
heart rate in beats / minute | 24 hours
  was measured before the block (0 min) and at 5, 10, 15, 30 min then 1, 2, 3, 6, 12,18and 24 h after the block.
peripheral oxygen saturation | 24 hours
  was measured before the block (0 min) and at 5, 10, 15, 30 min then 1, 2, 3, 6, 12,18and 24 h after the block.

CONTACTS AND LOCATIONS:
Locations (1):
- Zaher, Cairo, Egypt

REFERENCES:
- [Derived] Ghazaly HF, Aly AAA, Zaher ZZ, Hassan MM, Mahmoud AA. Comparison of the efficacy of two doses of dexmedetomidine as an adjunct to levobupivacaine in infraclavicular brachial plexus block: prospective double-blinded randomized controlled trial. BMC Anesthesiol. 2022 Nov 5;22(1):338. doi: 10.1186/s12871-022-01858-4. PMID 36335297